CLINICAL TRIAL: NCT02278731
Title: EFFECTS OF TWO EXERCISE PROTOCOLS IN POSTURAL BALANCE OF ELDERLY WOMEN
Brief Title: Exercise Protocols in Postural Balance Of Elderly Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual do PiauÍ (Other)
Responsible Party: Principal Investigator, Laiana Sepúlveda de Andrade Mesquita, UESPI, Universidade Estadual do PiauÍ
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U1111-1162-4778
Record Dates: First submitted 2014-10-22; First posted 2014-10-30 (Estimated); Last update posted 2014-10-30 (Estimated); Status verified 2014-10

CONDITIONS: Sarcopenia
Keywords: Physical activity; Rehabilitation; Older adults; Pilates; Proprioceptive neuromuscular facilitation
MeSH Terms: conditions — Sarcopenia; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control Group (No Intervention): The elderly in Control Group suffered no intervention and continued with their daily activities.
- Pilates Group (Active Comparator): Pilates group (PG), which underwent one-month (three times per week) training program with the Pilates method. This protocol consisted of Pilates exercises on the ground.Stretches were performed on upper trunk and lower limbs before the exercises. Subsequently, exercises that included the range of motion and strength of the upper limbs, trunk and lower limbs were performed, always associated with breathing and contraction of transversus abdominis muscles, in different positions, increasing repetitions and resistance in the weeks of the study, using the Swiss ball, thera-band and the magic circle.
  Interventions: Other: training program
- PNF Group (Active Comparator): PNF group that underwent one-month (three times per week) training program using the propriocptive neuromuscular facilitation method.The selected PNF diagonal patterns were chosen with all the basic procedures to the facilitation and according to three specific principles of PNF: rhythmic initiation, sustain and relax and reversal of antagonists. During the first week, one set of ten repetitions for each diagonal was performed; in the second week, two sets of ten repetitions and in the third and fourth weeks, three sets of ten repetitions were performed.
  Interventions: Other: training program

INTERVENTIONS:
Other: training program — Participants were randomly allocated to 1 of 3 groups: Pilates group (n=20), which underwent one-month (three times per week) training program with the Pilates method; PNF group (n=20), that underwent one-month (three times per week) training program using the PNF method; and Control group (n=18), that received no intervention during that one month and continued with their daily activities.
  Arms: PNF Group; Pilates Group

SUMMARY:
To determine and compare the effects of a training program with Pilates and Facilitation Neuromuscular Proprioceptive on balance and function in elderly women.

DETAILED DESCRIPTION:
Older women living in Teresina and participating in a local church project called "Pão dos Pobres" were randomly divided into three groups: Proprioceptive Neuromuscular Facilitation (PNFG), Pilates (PG) and Control(CG). Intervention: A training program (50 minutes session) was performed with the PNFG and the PG, 3 times a week, for 4 weeks. The elderly in CG suffered no intervention and continued with their daily activities. Main Outcome Measures: The stabilometric parameters, Berg Balance Scale score, functional reach test and Timed Up and Go test (TUG test) were measured before and one month after, in all participants.

ELIGIBILITY:
Inclusion Criteria:

* All the subjects were between 60 and 80 years old,
* sedentary and healthy

Exclusion Criteria:

-Orthopedic, cardiovascular, vestibular, psychological, neurological or any other impairment that would not allow the execution of all study tasks

Ages: 60 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2014-05; Primary Completion 2014-05 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Displacement of the center of pressure of the body | 1 month
  Displacement of the center of pressure of the body was collected using an electronic baropodometer, composed by a force platform with 1600 sensors. The subjects were oriented to be in a standing position in the platform, barefoot, bipedal support and with feet hip width apart.The kinetic variables related to body balance analyzed were: total displacement oscillation (TDO), amplitude of displacement of the center of pressure antero-posterior (ACPap), amplitude of displacement of the center of pressure medio-lateral (ACPml), displacement area (AREA), antero-posterior average speed (AAS), medio-lateral average speed (MAS) and total average speed (TAS).
Functional mobility on the Timed Up & Go test | 1 month
  The Timed Up & Go test (TUG) was applied to evaluate functional mobility involving speed, agility and dynamic balance of the elderly women, measuring the time in seconds spent by the volunteer to stand up from a chair (seat height 45 cm) without the help of arms, walk a three meters distance, turn around and return.
Static and dynamic balance on the Berg Balance test | 1 month
  The Berg Balance Scale consists in 14 tasks, on a 5-point ordinal scale, ranging from 0 (unable to perform the task) to 5 (performs the task independently). Scores of the 14 tasks are summed into a total score, ranging from 0 to 56 points, the highest score being related to better performance and values lower or equal to 45 points being related to prediction of falls.

REFERENCES:
- [Derived] Mesquita LS, de Carvalho FT, Freire LS, Neto OP, Zangaro RA. Effects of two exercise protocols on postural balance of elderly women: a randomized controlled trial. BMC Geriatr. 2015 Jun 2;15:61. doi: 10.1186/s12877-015-0059-3. PMID 26033080